CLINICAL TRIAL: NCT01283308
Title: The Diabetes Community Lifestyle Improvement Program (D-CLIP): A Translation Randomized Trial of a Culturally Specific Lifestyle Intervention for Diabetes Prevention in India
Brief Title: A Randomized Trial of Diabetes Prevention Through Lifestyle Change in India
Acronym: D-CLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Madras Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Venkat Narayan, Hubert Professor of Global Health and Epidemiology, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00016503; LT07-115 (Other: Other)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; India; Prevention & Control; Lifestyle Intervention; Translational Research
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Participants randomized to the standard of care group will receive standard lifestyle advice for diabetes prevention consistent with expert recommendations for a healthy lifestyle, including losing 5-10% of their excess body weight, following standard dietary recommendations to reduce calorie and fat intake, and exercising at least 150 minutes per week.
  Interventions: Behavioral: Standard of Care
- Lifestyle Intervention (Experimental): Intervention arm participants will participate in a step-wise model of diabetes prevention with the goal of reducing diabetes risk, primarily through (1) a weight loss of at least 7% and (2) 150 minutes or more per week of moderate level physical activity.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Intervention arm participants will attend 6 months of weekly classes where they will be taught the skills necessary to reach these goals. The curriculum for the classes is based on the DPP lesson plans. Social support will be provided by trained lay health educators and peer support groups. Participants who remain at highest risk of T2DM after four or more months in the program will be prescribed metformin in addition to continuing the lifestyle program. Metformin dosages will start at 500 mg per day, and, when appropriate, will increase to 1000 mg per day (given as 500 mg twice per day). This group will be comprised of individuals who have (1) Fasting plasma glucose values of 100 mg/dl or more and (2) elevated fasting HbA1c measures of 5.7% or more.
  Arms: Lifestyle Intervention
Behavioral: Standard of Care — Participants randomized to the standard of care group will meet with a physician and a dietician, attend one class/awareness lecture on diabetes prevention through weight loss and diet change and one class on exercise, and receive handouts reinforcing what they learn in class and with the dietician, fitness consultant, and physician.
  Arms: Standard of Care

SUMMARY:
People from the Indian subcontinent are more likely to get diabetes, even at younger ages. The Diabetes Community Lifestyle Improvement Program (D-CLIP) will test in a randomized trial if a culturally specific, community-based lifestyle and metformin (for individuals who do not respond to lifestyle change alone) intervention for men and women living in Chennai, India can effectively prevent type 2 diabetes in high-risk individuals. Lifestyle interventions are programs that seek to prevent disease by promoting changes in health behaviors, improved diet, increased physical activity, and weight loss. The results of this program will be used to make policy and public health recommendations, which will result in broader diabetes prevention efforts. The research team hypothesizes that this program will result in improvements in health (diabetes prevention, weight loss, and improvements in other markers of chronic disease) for intervention participants compared to participants in the control arm of the study.

DETAILED DESCRIPTION:
Aims: The Diabetes Community Lifestyle Improvement Program (D-CLIP) aims to implement and evaluate in a controlled, randomized trial the effectiveness, cost-effectiveness, and sustainability of a culturally appropriate, low-cost, and sustainable lifestyle intervention for the prevention of type 2 diabetes mellitus in India.

Methods: D-CLIP, a translational research project adapted from the methods and curriculum developed and tested for efficacy in the Diabetes Prevention Program, utilizes innovated methods (a step-wise model of diabetes prevention with lifestyle and metformin added when needed; inclusion of individuals with isolated impaired glucose tolerance, isolated impaired fasting glucose, and both; classes team-taught by professionals and trained community educators) with the goals of increasing diabetes prevention, community acceptability, and long-term dissemination and sustainability of the program. The primary outcome is, diabetes incidence, and secondary outcomes are cost-effectiveness, changes in anthropometric measures, plasma lipids, blood pressure, blood glucose, and HbA1c, and program acceptability and sustainability assessed using a mixed methods approach.

Conclusion: D-CLIP, a low-cost, community-based, research program, addresses the key components of translational research and can be used as a model for prevention of chronic diseases in other low- and middle-income country settings.

ELIGIBILITY:
Inclusion Criteria:

* Live in or near Chennai, India
* Aged 20-65 years
* A BMI >22 kg/m2 and/or a waist circumference >90 cm for men and >80 cm for women
* No prior diabetes diagnosis, except for gestational diabetes
* At high risk of developing diabetes (pre-diabetes) as defined by a casual capillary glucose greater than or equal to 110 (measured during screening) AND Baseline fasting glucose of 100-125 mg/dL and/or 2-hour post-load glucose of 140-199 mg/dL
* Willingness to consent to randomization

Exclusion Criteria:

* Does not fulfill inclusion criteria
* Currently pregnant or breastfeeding
* History of or biomarkers indicating heart disease, serious illness, cancer diagnosis in the past 5 years, or other conditions that may impede or prohibit participation in an unsupervised diet change and physical activity program.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2009-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Diabetes Incidence | Baseline through end of follow-up (mean follow-up time = 3 years)
  At baseline and follow-up visit(s), a 75-g oral glucose tolerance test will be administered to measure both 2-hour post-load glucose (2HG) and fasting plasma glucose (FPG). After the intervention and maintenance periods, blood glucose will be measured by a FPG test. Diabetes is diagnosed by a FPG≥126 mg/dL or a 2HG≥200 mg/dL. Diabetes incidence will be calculated by determining the proportion of individuals progressing from pre-diabetes to diabetes at each time point.

SECONDARY OUTCOMES:
Body Weight | Baseline through end of follow-up (mean follow-up time = 3 years)
  Weight will be measured in kilograms using a standardized, calibrated scale. Weight loss in kilograms and percent weight loss will be calculated.
Cost-effectiveness | Baseline through end of follow-up (mean follow-up time = 3 years)
  The cost-effectiveness of the intensive lifestyle program, from the perspectives of a single payer system and society, will be compared with standard lifestyle advice by conducting incremental cost-effective analyses in which the net costs and net effectiveness of the intensive lifestyle program and the standard lifestyle advice is calculated and expressed as a ratio.
Waist circumference | Baseline through end of follow-up (mean follow-up time = 3 years)
  Waist circumference in centimeters will be measured using a non-elastic tape measure. Change in waist circumference will be calculated.
Percent Body Fat | Baseline through end of follow-up (mean follow-up time = 3 years)
  Percent body fat will be measured using bioelectrical impedance (Beurer machine).
Blood Pressure | Baseline through end of follow-up (mean follow-up time = 3 years)
  Blood Pressure will be measured using standard procedures with an electronic BP apparatus.
Glycosylated hemoglobin (HbA1c) | Baseline through end of follow-up (mean follow-up time = 3 years)
  HbA1c will be measured from a fasting venous blood sample.
Plasma Lipids | Baseline through end of follow-up (mean follow-up time = 3 years)
  Plasma levels of high density lipoprotein (HDL), low density lipoprotein (LDL), triglycerides, and total cholesterol will be measured from fasting venous blood samples.
Beta Cell Function | Baseline through end of follow-up (mean follow-up time = 3 years)
  Changes in beta cell function [as measured by the Oral Disposition Index, calculated as (ΔI0-30 /ΔG0-30) x (1/fasting insulin)] and insulin resistance (using the Homeostasis Model Assessment of Insulin Resistance, HOMA-IR) will be calculated.
Dietary Intake | aseline through end of follow-up (mean follow-up time = 3 years)
  Changes in average diet are assessed by comparing the results of a 12-month food frequency questionnaire (FFQ) from baseline to the end of the intervention period and during follow-up.
Program Acceptability | Baseline through end of follow-up
  The acceptability of the intervention will be assessed through focus group discussions with participants who received the lifestyle intervention and phone interviews with program drop-outs.

CONTACTS AND LOCATIONS:
Overall Officials: Viswanathan Mohan, MD, PhD, Principal Investigator — Madras Diabetes Research Foundation/Dr. Mohan's Diabetes Specialities Centre; K.M. Venkat Narayan, MD, Principal Investigator — Emory University
Locations (1):
- Madras Diabetes Research Foundation, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Weber MB, Ranjani H, Anjana RM, Mohan V, Narayan KM, Gazmararian JA. Behavioral and psychosocial correlates of adiposity and healthy lifestyle in Asian Indians. Prim Care Diabetes. 2015 Dec;9(6):418-25. doi: 10.1016/j.pcd.2015.01.012. Epub 2015 Feb 26. PMID 25733342
- [Background] Staimez LR, Weber MB, Ranjani H, Ali MK, Echouffo-Tcheugui JB, Phillips LS, Mohan V, Narayan KM. Evidence of reduced beta-cell function in Asian Indians with mild dysglycemia. Diabetes Care. 2013 Sep;36(9):2772-8. doi: 10.2337/dc12-2290. Epub 2013 Apr 17. PMID 23596180
- [Background] Weber MB, Ranjani H, Meyers GC, Mohan V, Narayan KM. A model of translational research for diabetes prevention in low and middle-income countries: The Diabetes Community Lifestyle Improvement Program (D-CLIP) trial. Prim Care Diabetes. 2012 Apr;6(1):3-9. doi: 10.1016/j.pcd.2011.04.005. Epub 2011 May 26. PMID 21616737
- [Background] Ranjani H, Weber MB, Anjana RM, Lakshmi N, Narayan KMV, Mohan V. Recruitment challenges in a diabetes prevention trial in a low- and middle-income setting. Diabetes Res Clin Pract. 2015 Oct;110(1):51-59. doi: 10.1016/j.diabres.2015.07.013. Epub 2015 Aug 13. PMID 26321102
- [Background] Anjana RM, Ranjani H, Unnikrishnan R, Weber MB, Mohan V, Narayan KM. Exercise patterns and behaviour in Asian Indians: data from the baseline survey of the Diabetes Community Lifestyle Improvement Program (D-CLIP). Diabetes Res Clin Pract. 2015 Jan;107(1):77-84. doi: 10.1016/j.diabres.2014.09.053. Epub 2014 Oct 7. PMID 25458336
- [Result] Weber MB, Ranjani H, Staimez LR, Anjana RM, Ali MK, Narayan KM, Mohan V. The Stepwise Approach to Diabetes Prevention: Results From the D-CLIP Randomized Controlled Trial. Diabetes Care. 2016 Oct;39(10):1760-7. doi: 10.2337/dc16-1241. Epub 2016 Aug 8. PMID 27504014
- [Derived] Pyo E, Weber MB, Sivaram J, Staimez LR, Mohan V, Anjana RM, Haardorfer R, Ranjani H. Construct validity of the 12-item Short Form Health Survey (SF-12) version 2 and the impact of lifestyle modifications on the health-related quality of life among Indian adults with prediabetes: results from the D-CLIP trial. Qual Life Res. 2024 Jun;33(6):1593-1603. doi: 10.1007/s11136-024-03648-6. Epub 2024 Apr 12. PMID 38607494
- [Derived] Ford CN, Weber MB, Staimez LR, Anjana RM, Lakshmi K, Mohan V, Narayan KMV, Harish R. Dietary changes in a diabetes prevention intervention among people with prediabetes: the Diabetes Community Lifestyle Improvement Program trial. Acta Diabetol. 2019 Feb;56(2):197-209. doi: 10.1007/s00592-018-1249-1. Epub 2018 Nov 13. PMID 30426214
- [Derived] Cioffi CE, Ranjani H, Staimez LR, Anjana RM, Mohan V, Weber MB. Self-efficacy and diabetes prevention in overweight South Asians with pre-diabetes. BMJ Open Diabetes Res Care. 2018 Oct 15;6(1):e000561. doi: 10.1136/bmjdrc-2018-000561. eCollection 2018. PMID 30397491